CLINICAL TRIAL: NCT04617197
Title: Transcutaneous Electrical Nerve Stimulation With Frequency Specific Microcurrent Resonance Therapy for Non Specific Chronic Low Back Pain Patents: a Prospective Double Blinded, Randomized, Placebo Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Taiwan Resonant Waves Research Corp. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202009001
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Non Specific Chronic Low Back Pain
Keywords: Transcutaneous electrical nerve stimulation; non specific chronic low back pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Variable-frequency combination 1 (Experimental): Non disclosure
  Interventions: Device: Transcutaneous electrical nerve stimulation with frequency-specific microcurrent resonant therapy
- Variable-frequency combination 2 (Active Comparator): Non disclosure
  Interventions: Device: Transcutaneous electrical nerve stimulation with frequency-specific microcurrent resonant therapy
- Control (Placebo) (Placebo Comparator): Non-disclosure
  Interventions: Device: Transcutaneous electrical nerve stimulation with frequency-specific microcurrent resonant therapy

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation with frequency-specific microcurrent resonant therapy — Transcutaneous electrical nerve stimulation with frequency-specific microcurrent resonant therapy using (Dragon Waves Resonant Home Care Electronic Nerve Stimulator (DW-1330), Taiwan Resonance Wave Research Co., Taiwan R.O.C,)

SUMMARY:
Transcutaneous electrical nerve stimulation (TENS) is widely used for chronic pain. Recent studies showed frequency-specific microcurrent (FSM) resonant therapy was safe and effective in patients with non-specific chronic low back pain. However, there was no prospective, double-blinded randomized controlled trial to validate the clinical applicability. The goal of this trial is to verify safety and efficacy of FSM using a TENS device, Dragon Waves Resonant Home Care Electronic Nerve Stimulator-DW1330,(Taiwan Resonant Waves Research Co, Taiwan R.O.C), in 60 patients with non-specific low back pain.

DETAILED DESCRIPTION:
Several studies showed that frequency-specific microcurrent (FSM) resonance therapy delivered by transcutaneous electrical nerve stimulation (TENS) device is safe and effective in patients with non-specific low back pain. The regiment of variable-frequency combination (1-10000 Hz or 1-20000 Hz), continuous use for 36-60 mins per day and 30 to 180 days per session has been proven to be safe. To validate the clinical applicability of FSM by using a TENS device, DW-1330 (Taiwan Resonant Waves Research Co., Taiwan R.O.C.), a prospective, randomized, double-blinded trial is proposed. Investigators are going to recruit 60 patients with non-specific low back pain for at least 3 months. Clinical assessments include Numerical Rating Scale (NRS), Oswestry Disability Index (ODI), EuroQol instrument (EQ-5D), Pressure pain threshold (PPT), and Heart rate variability (HRV). The 60 patients were double-blinded, 1:1:1-randomly-distributed into 3 groups using different variable-frequency combinations: (1) Variable-frequency combination 1 (2) Variable-frequency combination 2 (3) Control(Placebo). During the surveillance period, a total of 2 visits and a telephone follow-up is set at Time point = 0, 2(telephone) and 4 week after recruitment. The primary endpoint is the change of NRS. The secondary endpoint is change of Heart rate variability (HRV). The safety evaluated index is the adverse event rate for all 3 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-80 years old, male or female.
2. Cases with normal psychological and communication functions who can cooperate with our study.
3. Cases who are willing to sign permits and cooperate with our study including follow up and examination.
4. Cases with complete clinical data and willing to accept investigation.

Exclusion Criteria:

1. Cases who diagnose pregnancy within 12 months before included.
2. Cases who diagnose with malignant disease.
3. Cases with a history of epilepsy.
4. Cases who diagnose with fracture without fixation.
5. Cases who diagnose with impaired sensation or psychological function.
6. Cases whose skin condition is not feasible to accept treatment.
7. Cases with pacemaker.
8. Cases who allergic to the conductive medium
9. Cases with a major psychiatric disorder such as schizophrenia or bipolar disorder.
10. Cases with severe visual or auditory disorder.
11. Cases who cannot communicate with the Mandarin language.
12. Other mental diseases are not suitable assessed by the PI

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Changes of non-specific chronic low back pain scaled by numerical rating scale | Time point = 0 week (before treatment), 2 week (during the treatment, by a telephone follow-up) and 4 week (after a 4-week treatment )
  In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity [1]. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.

SECONDARY OUTCOMES:
Changes of Heart rate variability | Time point = 0 week (before treatment) and 4 week (after a 4-week treatment )
  standard deviation of the normal-to-normal QRS interval (SDNN)

OTHER OUTCOMES:
Adverse rate | Time period during 4-week treatment
  Any adverse event accompany with the treatment will be document

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gozani SN. Fixed-site high-frequency transcutaneous electrical nerve stimulation for treatment of chronic low back and lower extremity pain. J Pain Res. 2016 Jun 28;9:469-79. doi: 10.2147/JPR.S111035. eCollection 2016. PMID 27418854
- [Result] Hazime FA, de Freitas DG, Monteiro RL, Maretto RL, Carvalho NA, Hasue RH, Joao SM. Analgesic efficacy of cerebral and peripheral electrical stimulation in chronic nonspecific low back pain: a randomized, double-blind, factorial clinical trial. BMC Musculoskelet Disord. 2015 Jan 31;16(1):7. doi: 10.1186/s12891-015-0461-1. PMID 25636503
- [Result] Gozani SN, Ferree TC, Moynihan M, Kong X. Impact of transcutaneous electrical nerve stimulation on sleep in chronic low back pain: a real-world retrospective cohort study. J Pain Res. 2019 Feb 25;12:743-752. doi: 10.2147/JPR.S196129. eCollection 2019. PMID 30881088